CLINICAL TRIAL: NCT05371392
Title: Polymorphism of the ITGA4 Gene (Integrin Subunit Alpha 4) in Chronic Lymphocytic Leukemia
Brief Title: Polymorphism of ITGA4 Gene in Chronic Lymphocytic Leukemia
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amer Ahmed Youssef Abdalkareem, Specialist of clinical and chemical pathology, Sohag University
Other Study IDs: soh-med-22-04-21
Record Dates: First submitted 2022-04-29; First posted 2022-05-12 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient group
- control group

SUMMARY:
Chronic lymphocytic leukemia (CLL) is a clonal lymphoproliferative disorder that is characterized by heterogeneous presentation at the clinical and molecular levels. ITGA4 protein has been found to be deregulated in CLL with adverse clinical outcome. ITGA4 gene (CD49d) encodes a member of the integrin alpha chain family of proteins and is considered a negative prognosticator in CLL with aggressive course and short time to treatment.

The aim of the study:

is to investigate ITGA4 gene expression pattern in CLL.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed CLL.

Exclusion Criteria:

* ▪ Patients previously diagnosed as CLL and received treatment before.

  * Patients with other solid tumors.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: newly diagnosed patients with Chronic lymphocytic leukemia
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
ITGA4 gene expression pattern in chronic lymphocytic leukemia | 1 year following the startpoint of the study
  Detection of ITGA4 gene expression in blood samples in patients with chronic lymphocytic leukemia, Briefly, total RNA and genomic DNA extraction from fresh peripheral blood samples by Real-time -RT-polymerase chain reaction system (RT-PCR) will be carried out. Rate of ITGA4 gene expression will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Amer Ahmed Youssif, Principal Investigator — Sohag University
Locations (1):
- Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided